CLINICAL TRIAL: NCT03435471
Title: Does the Use of Clinician Directed Prophylactic Swallowing Therapy in Patients Undergoing Definitive Chemoradiation for Head and Neck Cancer Improve Swallowing Function Outcomes?
Brief Title: Outcomes of Prophylactic Swallowing Therapy in Patients Undergoing Definitive Chemoradiation for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Donna S. Lundy, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180084
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Head and Neck Cancer; Oropharynx Cancer
Keywords: Prophylactic Swallowing Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G1 - Clinician-Directed Therapy (Experimental): Clinician-Directed Weekly Swallowing Therapy: Once weekly face-to-face meetings with a study speech pathologist for a total of six sessions, to participate in active swallowing exercises and review the home swallowing exercise program. Each session will last 30 minutes +/- ten minutes. Other assessments include:
  * Clinician-Directed Prophylactic Swallowing Exercises
  * Prophylactic Swallowing Home Exercise Program
  * Penetration/Aspiration Scale (PAS)
  * Functional Oral Intake Scale (FOIS)
  * Eating Assessment Tool-10 (EAT-10)
  * University of Washington Quality of Life (UW-QOL)
  * Performance Status Scale for Head and Neck Cancer Patients (PSS-HN)
  * DIGEST Safety Grade
  Interventions: Other: Prophylactic Swallowing Home Exercise Program; Other: Clinician-Directed Prophylactic Swallowing Exercises
- G2 - Patient-Directed Home Therapy (Active Comparator): Patient-Directed Home Swallowing Therapy: One face-to-face meeting with a study speech pathologist prior to initiation of treatment. During that session, they will be encouraged to practice the given exercises independently on a specific daily schedule regime throughout their treatment. Other assessments include:
  * Prophylactic Swallowing Home Exercise Program
  * Penetration/Aspiration Scale (PAS)
  * Functional Oral Intake Scale (FOIS)
  * Eating Assessment Tool-10 (EAT-10)
  * University of Washington Quality of Life (UW-QOL)
  * Performance Status Scale for Head and Neck Cancer Patients (PSS-HN)
  * DIGEST Safety Grade
  Interventions: Other: Prophylactic Swallowing Home Exercise Program

INTERVENTIONS:
Other: Prophylactic Swallowing Home Exercise Program — The home exercise program will consist of six exercises that are recommended to be practiced three times per day. Subjects will complete a weekly exercise log to track compliance.
Other: Clinician-Directed Prophylactic Swallowing Exercises — Once weekly face-to-face meetings with a study speech pathologist for a total of six sessions, to participate in active swallowing exercises
  Arms: G1 - Clinician-Directed Therapy

SUMMARY:
Clinician directed prophylactic swallowing therapy will improve immediate (four weeks +/- two weeks) and short-term (26 weeks +/- four weeks) post-treatment swallowing function and quality of life versus patient directed home exercises.

The purpose of this prospective, interventional, pilot investigation is to determine whether clinician directed swallowing therapy will improve patient swallowing function outcomes and quality of life in the immediate and short-term basis compared to patients receiving standard of care patient directed independent home swallowing therapy. Patient compliance with home exercises programs is reportedly inconsistent. Patients may experience changes in their physical functioning and overall well-being that may impact their ability to follow-through with independent home therapy. Clinician directed swallowing therapy allows for ongoing assessment of changes that may warrant modifying the therapy program in terms of intensity of exercises and/or expectations. This facilitates individualizing the patient's therapy plan to maximize their function and ability to achieve goals. It is anticipated that individualizing swallowing therapy through weekly session will result in improved swallowing function.

DETAILED DESCRIPTION:
This is a single-site, two-arm, 1:1 randomized, prospective, interventional, pilot study to determine whether clinician directed swallowing therapy will improve patient swallowing function outcomes when compared to patient-directed home-based swallowing therapy.

The investigators anticipate at least 40 subjects will need to be enrolled/consented in order to obtain the accrual goal of 15 evaluable subjects for each group for a total of 30 participants.

All subjects in each group will receive a face-to-face education session with a speech pathologist to review a recommended program of swallowing exercises prior to initiation of chemoradiation at their baseline (pre-treatment evaluation session).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of head and neck cancer (sites: oropharynx: human papillomavirus (HPV) related and non HPV related tonsil and base of tongue)
2. Scheduled to undergo definitive chemoradiation therapy
3. At least 18 years of age or older
4. Subject must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Surgical management in addition to chemoradiation therapy;
2. Cancer of the sinus, brain, or parotid;
3. Prior treatment for head and neck cancer;
4. Receiving chemoradiation treatment at an outside institution (i.e., non-University of Miami (UM) clinic);
5. Prior history of dysphagia unrelated to the current diagnosis of head and neck cancer;
6. Prior neurologic disorder (i.e., Cerebrovascular accident (CVA), Traumatic brain injury (TBI), dementia) or current degenerative neuromuscular disease;
7. History of prior c-spine surgery;
8. History of prior vocal fold immobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Change in swallowing status | Baseline, Up to 6 weeks
  Swallowing status will be measured using Functional Oral Intake Scale (FOIS). FOIS has a range from 0 (most restrictive) to 7 (least restrictive).

SECONDARY OUTCOMES:
Change in swallowing status as measured by FOIS | Baseline, Up to 30 weeks
  FOIS has a range from 0 (most restrictive) to 7 (least restrictive).
Change in quality of life as measured by PSS-HN | Baseline to 6 weeks, Baseline to 30 weeks
  Performance Status Scale - Head and Neck (PSS-HSN) is a questionnaire with a total score ranging from 100 (normal function) to 0 (limited function).
Change in quality of life as measured by EAT-10 | Baseline to 6 weeks, Baseline to 30 weeks
  Eating Assessment Tool-10 (EAT-10) is a questionnaire with a total score ranging from 0 to 40 with the lower score indicating better function.
Change in quality of life as measured by UW-QOL | Baseline to 6 weeks, Baseline to 30 weeks
  University of Washington Quality of Life (UW-QOL) is a questionnaire with a total score ranging from 0 to 100 with the higher score indicating poorer health outcomes.
Proportion of patients requiring further swallowing therapy | Baseline to 6 weeks, Baseline to 30 weeks
  Proportion of patients requiring further swallowing therapy post study intervention as per treating physician discretion
Change in Pharyngeal Swallowing Efficiency and Safety as measured by DIGEST Safety Grade | Baseline to 6 weeks, Baseline to 30 weeks
  DIGEST is a measure of pharyngeal swallowing efficiency and safety. The DIGEST measure incorporates 2 measures:
  1. Safety as determined by the Penetration Aspiration Scale with a score ranging from 0 (safe) to 4 (life-threatening unsafe); and
  2. Efficiency as determined by the quantity of residue observed on the videoflouroscopic swallowing study with a score ranging from 0 (efficient) to 4 (life-threatening inefficiency).
  These two measures combine for an overall score, ranging from 0 (no pharyngeal dysphagia) to 4 (life-threatening dysphagia).

CONTACTS AND LOCATIONS:
Overall Officials: Donna S Lundy, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No